CLINICAL TRIAL: NCT00645008
Title: Stressors Associated With Cardiac Surgery Intensive Care Treatment
Brief Title: Identification of Dominate Stressors in the Intensive Care Unit (ICU)
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0801009626
Record Dates: First submitted 2008-03-19; First posted 2008-03-27 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Cardiac Surgery Intensive Care Treatment
Keywords: Stressors; Patient Satisfaction; Cardiothoracic-Intensive Care Unit; Coronary bypass patient
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Undergoing cardiopulmonary bypass surgery and the subsequent admission to the intensive care unit (ICU) is known to be a stressful event to the patient. As patients prepare for open-heart surgery it is natural for them to feel anxious and concerned about all the various procedures involved in the process. Members of both the surgical and anesthesia team explain the purpose of each procedure and all issues associated with the procedures in great detail in order to better prepare the patient, ease their anxiety and aid their recovery.

The underlying assumption for past investigations into overall patient satisfaction has been that the stressors inherent in the experience of illness and hospitalization have an adverse effect on patient recovery and can possibly prolong the recuperative process. Previous studies have shown that the specific performance of a team in regard to the effects of the stressors on the patient's status is key to providing optimal patient care in the ICU environment. Since the ICU stay is a difficult experience in the life of a patient, stressor predictability might allow for better physical and psychological conditions for the patient's recovery.

Although there is a myriad of published research available on the potential stressors related to an ICU stay, there is a dearth of investigation into the inherently more intense circumstances surrounding a stay in the Cardiothoracic Intensive Care Unit (CT-ICU). By examining the stressors in the CT-ICU changes can be made by the medical care team and/or hospital that can ultimately enhance the patient experience in the CT-ICU.

The purpose of this study is to reduce or completely eliminate stressors present in the CT-ICU as identified by the cardiac bypass patient. Identification of events and conditions considered stressful in the ICU will allow the professional team to determine which stressors are amendable to intervention and tailor patient care accordingly.

DETAILED DESCRIPTION:
Hypothesis: Identification of events and conditions considered stressful by the cardiopulmonary bypass patient would allow the professional team to determine which stressors are amendable to intervention and tailor patient care accordingly in order to improve future patient care experience in the intensive care unit.

Research Question: What are the dominant stressors associated with intensive care treatment as perceived by the patient, and what measures can be taken by the professional team members of the unit to decrease or eliminate these stressors entirely?

Purpose: The purpose of this study is to reduce or completely eliminate stressors present in the CT-ICU as identified by the coronary bypass patient. Identification of events and conditions considered stressful in the ICU will allow the professional team to determine which stressors are amendable to intervention and tailor patient care accordingly.

Design: Analytical survey

Protocol: Patients will be selected based on admission to the ICU following cardiopulmonary bypass surgery. We plan to survey 160 patients in order to identify the main stressors in the ICU as perceived by the patient themselves. A study investigator will enroll subjects after obtaining oral informed consent. We plan to approach eligible candidates once they have been discharged from the ICU to the step-down unit (4C). Subjects will be asked to complete a short questionnaire that will ask them to assess stressors associated with their stay in the CT-ICU. Preliminary analysis will be done to appraise the leading stressors after enrolling 80 patients in the study. Once dominate stressors have been identified, we will conduct several in-services in order to educate the CT-ICU team members of the amendable stressors. We will then enroll another 80 patients in order to evaluate whether or not the stressors have been reduced and/or eliminated.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the ICU following cardiopulmonary bypass surgery (AVR/MVR and/or CABG)
* Conscious, alert and having the capacity to consent and answer survey questions, i.e. no dementia
* Adults > 18 years old

Exclusion Criteria:

* Admitted to the CT-ICU for greater than 4 days (>96 hours)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study involves patients both male and female who are admitted to the intensive care unit immediately following cardiopulmonary bypass for either myocardial revascularization or valvular surgery.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Identification of stressors present in the CT-ICU (as recognized by completed surveys) | Analysis after completion of 80 surveys

SECONDARY OUTCOMES:
Reduction and/or elimination of dominate stressors present in the CT-ICU | Analysis after completion of 160 surveys

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Kerr, MD, MBA, Principal Investigator — The NewYork-Presbyterian Hospital-Weill Cornell Medical College
Locations (1):
- The NewYork-Presbyterian Hospital-Weill Cornell Medical College, Cardiothoracic Intensive Care Unit (4W) - NYPH, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Will not be shared